CLINICAL TRIAL: NCT06561464
Title: Reflections of Oxygen Delivery Methods Applied in Acute Exacerbations of Chronic Obstructive Pulmonary Disease (COPD) on Blood Gas and Spirometer Measurements
Brief Title: Evaluation of Oxygen Delivery Methods in Acute Exacerbations of Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Emine Sarcan, Doctor, Ankara Etlik City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ES-COPD
Record Dates: First submitted 2024-07-08; First posted 2024-08-20 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Chronic Obstructive Pulmonary Disease Exacerbation
Keywords: Non-invasive ventilation; EzPAP®; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: EzPAP® will be applied (Active Comparator): This group, selected randomly and allocated to non-invasive ventilation (NIV) indication, will receive EzPAP® as a single-blind randomized trial.
  Non-Invasive Indications for Acute Exacerbations of COPD:
  (At least two of the following parameters must be present)
  * Moderate to severe dyspnea leading to the use of accessory respiratory muscles and paradoxical abdominal movements,
  * Tachypnea (respiratory rate > 25 breaths per minute),
  * Arterial blood gas (ABG) results with pH < 7.35, pCO2 > 45 mmHg, or
  * PaO2/FiO2 < 200 mmHg
  Interventions: Device: EzPAP®
- Group B: NIMV will be applied. (Active Comparator): This group, selected randomly and allocated to non-invasive ventilation (NIMV) as a single-blind randomized trial, NIMV provides respiratory support during both expiration and inspiration with either continuous positive airway pressure (CPAP) or bi-level positive airway pressure (BiPAP), which operates with intermittent positive pressure.
  Non-Invasive Indications for Acute Exacerbations of COPD:
  (At least two of the following parameters must be present)
  * Moderate to severe dyspnea leading to the use of accessory respiratory muscles and paradoxical abdominal movements,
  * Tachypnea (respiratory rate > 25 breaths per minute),
  * Arterial blood gas (ABG) results with pH < 7.35, pCO2 > 45 mmHg, or
  * PaO2/FiO2 < 200 mmHg
  Interventions: Device: Non-invasive mechanical ventilation (NIMV)

INTERVENTIONS:
Device: EzPAP® — EzPAP® is a portable, single-use respiratory exercise device that provides positive expiratory pressure during expiration while supporting respiration during inspiration. Its use has been increasing in recent years as an oxygenation device. It is portable, single-use, easy to use, well-tolerated, and cost-effective. EzPAP® helps increase functional capacity in the lungs and reduces atelectasis. With EzPAP®, an oxygen flow of 5-8 L/min reaches the patient as 35-42% fractionated oxygen, thus quadrupling the oxygen flow.
  Arms: Group A: EzPAP® will be applied
Device: Non-invasive mechanical ventilation (NIMV) — NIMV provides respiratory support during both expiration and inspiration through continuous positive airway pressure (CPAP) or bi-level positive airway pressure (BiPAP). Treatment success can be monitored within the first 2 hours by the improvement in oxygenation and reduction in pCO2 levels
  Arms: Group B: NIMV will be applied.

SUMMARY:
To examine the effects of oxygen therapy methods applied as indicated in COPD acute exacerbations on blood gas results and spirometric measurements.

DETAILED DESCRIPTION:
Patients requiring non-invasive ventilation will be divided into two groups: one group will receive NIMV in the form of Continuous Positive Airway Pressure (CPAP) or Bi-level Positive Airway Pressure (BiPAP). The other group will receive EzPAP® (a non-invasive positive airway pressure device). For both groups, blood gas results and hand-held spirometer parameters, including Forced Vital Capacity (FVC), Peak Expiratory Flow (PEF), and Forced Expiratory Volume in one second (FEV1), will be evaluated before and after the application.It is aimed to evaluate the effect of COPD noninvasive treatment methods on hospitalization and mortality processes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute exacerbation of COPD,
* Those without a history of trauma,
* Patients who have not undergone any lung surgery previously,
* Patients capable of providing written and verbal consent.

Exclusion Criteria:

* Patients without acute exacerbation of COPD,
* Pregnancy, suspected pregnancy,
* Those who have undergone any lung surgery previously,
* Patients with a history of trauma,
* Intubated patients and those not compliant with treatments,
* Patients unable to provide written and verbal consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Arterial blood gas and spirometry values will be examined before and after treatment administration to patients. | Patients will receive 2-hour treatment (EzPAP and NIMV) and then measurements will be taken 30 minutes after the completion of treatment in both groups.
  Patients meeting the inclusion criteria will be enrolled in the study after obtaining informed consent.
  1. Before treatment, the following parameters will be assessed:
     * Blood pressure (mmHg)
     * Oxygen Saturation (%)
     * Respiratory rate /min,
     * Heart rate/min
     * pH
     * pCO2-mmHg
     * PaO2-mmHg
     * HCO3-mEq/L
     * Lactate-mmol/L
     * FEV1-Liter
     * FVC-Liter
     * - PEF-L/min
  2. After treatment, the following parameters will be assessed:
     * Blood pressure (mmHg)
     * Oxygen Saturation (%)
     * Respiratory rate /min,
     * Heart rate/min
     * pH
     * pCO2-mmHg
     * PaO2-mmHg
     * HCO3-mEq/L
     * Lactate-mmol/L
     * FEV1-Liter
     * FVC-Liter
     * PEF-L/min
Evaluation of the patient's mortalite after treatment. | The 30-day mortality of the patients will be evaluated.
  - 30-day mortality of the patients will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Burak Erdem, Study Director — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
A decision will be made after the study is written up as an article.

REFERENCES:
- [Background] Iberl G, Bornitz F, Schellenberg M, Wiebel M, Herth FJ, Kreuter M. [Respiratory therapy with Ez-PAP for treatment of dynamic hyperinflation in patients with severe COPD and emphysema]. Pneumologie. 2014 Sep;68(9):604-12. doi: 10.1055/s-0034-1377483. Epub 2014 Sep 9. German. PMID 25203820
- [Background] Rieg AD, Stoppe C, Rossaint R, Coburn M, Hein M, Schalte G. [EzPAP(R) therapy of postoperative hypoxemia in the recovery room : experiences with the new compact system of end-expiratory positive airway pressure]. Anaesthesist. 2012 Oct;61(10):867-74. doi: 10.1007/s00101-012-2083-4. Epub 2012 Sep 27. German. PMID 23011043
- [Derived] Sarcan E, Erdem AB, Yazla M, Uysal SB, Celikel E. Comparison of positive expiratory pressure device versus non-invasive ventilation on outcomes in acute exacerbation of chronic obstructive pulmonary disease in the emergency department. BMC Emerg Med. 2025 Jul 1;25(1):110. doi: 10.1186/s12873-025-01267-z. PMID 40596843